CLINICAL TRIAL: NCT06758947
Title: Upadacetinib Versus MMF in SSc-ILD
Brief Title: Use of Selective JAK Inhibitor in ILD and Skin Tightness of Systemic Sclerosis Versus MMF
Acronym: upadacetinib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Professor of Rheumatology, faculty of medicine Assuit university, Egypt, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Upadacetinib in SscILD; Assuit university (Other: Assuit university)
Record Dates: First submitted 2024-12-21; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Interstitial Lung Disease Due to Systemic Disease (Disorder)
Keywords: ILD
MeSH Terms: interventions — upadacitinib

STUDY DESIGN:
Intervention Model Description: Randomised double blinded clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- upadacitinib (Experimental): upadacitinib 15 mg oral once daily
  Interventions: Drug: Upadacitinib 15 MG
- MMF (Active Comparator): MMF 2 gm oral daily
  Interventions: Device: Cellcept Oral Product

INTERVENTIONS:
Drug: Upadacitinib 15 MG — oral tablet upadacitinib
  Other Names: Upadacitinib
  Arms: upadacitinib
Device: Cellcept Oral Product — active control group 2000mg MMF daily
  Other Names: MMF
  Arms: MMF

SUMMARY:
Systemic sclerosis (SSc) is a systemic autoimmune disease with heterogeneous clinical presentation and prognosis. JAK inhibitors reduced cutaneous and pulmonary fibrosis in mice models of SSc. Clinical data regarding the efficacy and safety of JAK inhibitors in SSc patients are scarce

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a systemic autoimmune disease with heterogeneous clinical presentation and prognosis. JAK inhibitors reduced cutaneous and pulmonary fibrosis in mice models of SSc. Clinical data regarding the efficacy and safety of JAK inhibitors in SSc patients are scarce. Upadacitinib mechanism of action JAK-STAT pathways are composed of four JAK kinases and seven STATs (STAT1-6, including homologs STAT5a and STAT5b). A cytokine binding to its receptor initiates the signaling cascade as well as the subsequent association/rearrangement of the receptor subunits. This rearrangement enables JAK activation by transphosphorylation and, upon activation, JAKs phosphorylate the receptors.

ELIGIBILITY:
Inclusion Criteria:

* all patients are systemic sclerosis disease duration more than 3 years limited and diffuse types ground glass at HRCT DLCO< 80% decline in FVC >10% in last 12months

Exclusion Criteria:

* associated other CT diseases disease duration < 3 years kidney disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
forced vital capacity | 52 week
  FVC reduction of 15%

SECONDARY OUTCOMES:
High resolution chest computed tomography | 52 week
  HRCT chest pattern changes ground glass appearance
modefided Rodnan skin score | 52 week
  skin score for tightness grade more than 14 is worse

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hassanien, professor, Principal Investigator — Assiut University
Locations (1):
- Medicinr, Asyut, Alabama, Egypt

IPD SHARING:
Plan to Share IPD: Yes
allocation to which study arm and the outcome data analysis
Supporting Information: Study Protocol
Time Frame: 15 july 2025